CLINICAL TRIAL: NCT00005298
Title: Inflammation, Autonomic Dysfunction and Airway Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 2021; R01HL045089 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-06

CONDITIONS: Lung Diseases; Asthma; Bronchitis; Inflammation
MeSH Terms: conditions — Lung Diseases; Asthma; Bronchitis; Inflammation

SUMMARY:
To determine whether airway inflammation secondary to inhalation of specific allergens and other environmental agents and functional imbalance of the autonomic nervous system played important roles in asthma and chronic bronchitis.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma and chronic bronchitis are among the most common chronic diseases afflicting middle-aged and elderly adults in the United States, respectively occurring in 4 percent and 5 percent of the population in these age groups. While chronic bronchitis is often caused by cigarette smoking and asthma often occurs in nonsmokers in association with atopy, the two conditions may be difficult to differentiate in many middle-aged and older adults and may share a number of pathophysiologic features including increased airway smooth muscle tone, increased airway responsiveness to bronchoconstricting stimuli, and bronchial mucus hypersecretion. The precise mechanisms which produce the alterations of airway function are not clear. Such functional alterations may be caused by airway inflammation and abnormalities of the autonomic nervous system; however, there are little population data available regarding the importance of airway inflammation and disordered neural regulation in the pathogenesis of airway hyperresponsiveness and mucus hypersecretion. Also, little is known about potential interactions between airway inflammation and disordered neural regulation of airway function in the pathogenesis of chronic airways disease. Information on the relationships may offer insights into the pathophysiologic mechanisms underlying asthma and chronic bronchitis in adults.

DESIGN NARRATIVE:

The study was cross-sectional and used a subgroup of the Normative Aging Study, a longitudinal study of aging in men established by the Veterans Administration in 1963. The study used data normally collected during NAS examinations and included smoking history, socio-economic status, anthropometry, respiratory symptoms and illnesses, and pulmonary function. New data were collected on: indices of inflammation as indicated by histamine, leukotriene, and serotonin in urine; autonomic activity as indicated by urinary catecholamine excretion and heart rate variation induced by deep breathing; autonomic responsiveness as measured by pupillary alpha-adrenergic and cholinergic responses.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-07; Study Completion 1993-06 (Actual)

REFERENCES:
- [Background] Lazarus R, Sparrow D, Weiss ST. Effects of obesity and fat distribution on ventilatory function: the normative aging study. Chest. 1997 Apr;111(4):891-8. doi: 10.1378/chest.111.4.891. PMID 9106566
- [Background] Sparrow D, O'Connor GT, Weiss ST, DeMolles D, Ingram RH Jr. Volume history effects and airway responsiveness in middle-aged and older men. The Normative Aging Study. Am J Respir Crit Care Med. 1997 Mar;155(3):888-92. doi: 10.1164/ajrccm.155.3.9117022.
- [Background] Shadick NA, Sparrow D, O'Connor GT, DeMolles D, Weiss ST. Relationship of serum IgE concentration to level and rate of decline of pulmonary function: the Normative Aging Study. Thorax. 1996 Aug;51(8):787-92. doi: 10.1136/thx.51.8.787. PMID 8795665
- [Background] Sparrow D, O'Connor GT, Young JB, Rosner B, Weiss ST. Relationship of urinary serotonin excretion to cigarette smoking and respiratory symptoms. The Normative Aging Study. Chest. 1992 Apr;101(4):976-80. doi: 10.1378/chest.101.4.976. PMID 1372851
- [Background] Freeman R, Weiss ST, Roberts M, Zbikowski SM, Sparrow D. The relationship between heart rate variability and measures of body habitus. Clin Auton Res. 1995 Oct;5(5):261-6. doi: 10.1007/BF01818890. PMID 8563458
- [Background] O'Connor GT, Sparrow D, Weiss ST. A prospective longitudinal study of methacholine airway responsiveness as a predictor of pulmonary-function decline: the Normative Aging Study. Am J Respir Crit Care Med. 1995 Jul;152(1):87-92. doi: 10.1164/ajrccm.152.1.7599868.
- [Background] Annema JT, Sparrow D, O'Connor GT, Rijcken B, Koeter GH, Postma DS, Weiss ST. Chronic respiratory symptoms and airway responsiveness to methacholine are associated with eosinophilia in older men: the Normative Aging Study. Eur Respir J. 1995 Jan;8(1):62-9. doi: 10.1183/09031936.95.08010062. PMID 7744195
- [Background] Kawachi I, Sparrow D, Vokonas PS, Weiss ST. Decreased heart rate variability in men with phobic anxiety (data from the Normative Aging Study). Am J Cardiol. 1995 May 1;75(14):882-5. doi: 10.1016/s0002-9149(99)80680-8. PMID 7732994
- [Background] Ward KD, Sparrow D, Vokonas PS, Willett WC, Landsberg L, Weiss ST. The relationships of abdominal obesity, hyperinsulinemia and saturated fat intake to serum lipid levels: the Normative Aging Study. Int J Obes Relat Metab Disord. 1994 Mar;18(3):137-44. PMID 8186810
- [Background] Ward KD, Sparrow D, Landsberg L, Young JB, Vokonas PS, Weiss ST. The relationship of epinephrine excretion to serum lipid levels: the Normative Aging Study. Metabolism. 1994 Apr;43(4):509-13. doi: 10.1016/0026-0495(94)90085-x. PMID 8159112
- [Background] O'Connor GT, Sparrow D, Weiss ST. Normal range of methacholine responsiveness in relation to prechallenge pulmonary function. The Normative Aging Study. Chest. 1994 Mar;105(3):661-6. doi: 10.1378/chest.105.3.661. PMID 8131522
- [Background] Sparrow D, O'Connor GT, Rosner B, Weiss ST. Predictors of longitudinal change in methacholine airway responsiveness among middle-aged and older men: the Normative Aging Study. Am J Respir Crit Care Med. 1994 Feb;149(2 Pt 1):376-81. doi: 10.1164/ajrccm.149.2.8306033.
- [Background] Weiss ST, Sparrow D, O'Connor GT. The interrelationship among allergy, airways responsiveness, and asthma. J Asthma. 1993;30(5):329-49. doi: 10.3109/02770909309056738. No abstract available. PMID 8407734
- [Background] Sparrow D, O'Connor GT, Rosner B, DeMolles D, Weiss ST. A longitudinal study of plasma cortisol concentration and pulmonary function decline in men. The Normative Aging Study. Am Rev Respir Dis. 1993 Jun;147(6 Pt 1):1345-8. doi: 10.1164/ajrccm/147.6_Pt_1.1345. PMID 8503543
- [Background] Ohman JL Jr, Sparrow D, MacDonald MR. New onset wheezing in an older male population: evidence of allergen sensitization in a longitudinal study. Results of the normative aging study. J Allergy Clin Immunol. 1993 Mar;91(3):752-7. doi: 10.1016/0091-6749(93)90195-l. PMID 8454798
- [Background] O'Connor GT, Sparrow D, Segal M, Weiss ST. Risk factors for ventilatory impairment among middle-aged and elderly men. The Normative Aging Study. Chest. 1993 Feb;103(2):376-82. doi: 10.1378/chest.103.2.376. PMID 8432122
- [Background] Sparrow D, O'Connor GT, Basner RC, Rosner B, Weiss ST. Predictors of the new onset of wheezing among middle-aged and older men. The Normative Aging Study. Am Rev Respir Dis. 1993 Feb;147(2):367-71. doi: 10.1164/ajrccm/147.2.367. PMID 8430960